CLINICAL TRIAL: NCT06767137
Title: Comparative Efficacy of Bedtime Restriction Therapy and Cognitive Behavioral Therapy for Insomnia - a Randomized Controlled Non-inferiority Trial
Brief Title: Comparative Efficacy of BRT and CBT-I for Insomnia
Acronym: SLEEPwindow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Nissen (Other)
Responsible Party: Sponsor-Investigator, Christoph Nissen, Prof. Dr. med., University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-01324
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Insomnia Disorders; Insomnia Disorder; Insomnia; Insomnia Chronic; Insomnia, Primary; Insomnia, Nonorganic; Insomnia Type; Sleep Disorder
Keywords: insomnia; cognitive behavioral therapy; bedtime restriction; sleep restriction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive behavioral therapy for insomnia (CBT-I) (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBT-I)
- Bedtime restriction (BRT) (Experimental)
  Interventions: Behavioral: Bedtime restriction (BRT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia (CBT-I) — Cognitive Behavioral Therapy for Insomnia (CBT-I) is a gold-standard, evidence-based treatment combining techniques to improve the clinical symptomatology of insomnia. Delivered in six 90-minute group sessions over six weeks, it includes: sleep education (i.e. understanding sleep mechanisms and influencing factors), bedtime restriction (i.e. aligning bedtimes with reported sleep duration), stimulus control (i.e. getting out of bed when unable to sleep), cognitive therapy (i.e. addressing dysfunctional sleep beliefs), relaxation techniques (i.e. using methods like progressive muscle relaxation).
  Arms: Cognitive behavioral therapy for insomnia (CBT-I)
Behavioral: Bedtime restriction (BRT) — Bedtime Restriction Therapy (BRT): A behavioral intervention aimed at improving the clinical symptomatology of insomnia by aligning time spent in bed with reported sleep duration. Participants attend four 60-minute group therapy sessions over six weeks. The intervention includes: setting individualized sleep windows based on sleep diaries, regular adjustment of sleep schedules to enhance sleep pressure, group discussions to address implementation challenges and maintain motivation.
  BRT focuses exclusively on bed time restriction without additional cognitive or relaxation components, making it a simplified, resource-efficient approach to treating insomnia.
  Arms: Bedtime restriction (BRT)

SUMMARY:
This study evaluates two behavioral treatments for patients with insomnia disorder: Bedtime Restriction Therapy (BRT) and Cognitive Behavioral Therapy for Insomnia (CBT-I). Both therapies aim to improve the clinical symptomatology of insomnia by teaching participants techniques to better manage their sleep schedule and habits. BRT is a simpler and shorter therapy focused on aligning the time spent in bed with reported sleep time. CBT-I includes additional components such as relaxation techniques and cognitive exercises. The study will compare these treatments to see if BRT is as effective as CBT-I in improving the clinical symptomatology of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-5 criteria for insomnia disorder.
* Adults aged 18 to 80 years
* Capable of giving written informed consent.
* Sufficient fluency in the study site's language (i.e., German or French) to understand all study-related information.

Exclusion Criteria:

* Unstable, progressive, or degenerative medical condition
* Acute pain or poorly managed chronic pain
* Suicidality
* Uncontrolled psychiatric condition requiring treatment outside of study
* Alcohol or drug abuse or dependency
* Diagnosis of psychosis, bipolar disorder, autism, borderline personality disorder, or antisocial personality disorder
* Clinical evidence of sleep disorders other than insomnia (e.g., sleep apnea, restless legs, periodic limb movements in sleep, parasomnia)
* Evidence of intellectual disability
* Regular intake of benzodiazepines (BZD) or benzodiazepine receptor agonists (BZDRA)
* Alteration of medication within 4 weeks prior to study treatment or planned alteration during the trial period (stable medication except BZD or BZDRA does not lead to exclusion)
* Current other psychotherapy for insomnia
* Known pregnancy or breastfeeding
* Inability to comply with study procedure
* Insufficient fluency in German or French to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) summary scores | Baseline (T0) to 6 weeks (T1), 3 months (T2), and 6 months (T3)

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Universität Bern, Psychotherapeutische Praxisstelle, Bern, Canton of Bern
  - Service des specialités psychiatriques, Hôpitaux universitaires de Genève, Geneva, Canton of Geneva

IPD SHARING:
Plan to Share IPD: No